CLINICAL TRIAL: NCT05766059
Title: Novel Non-invasive Brain Stimulation Techniques in Neurological Rehabilitation: Cross-modal Paired Associative Stimulation (PAS) Protocols to Promote Plastic Reorganization in Stroke and Phantom Limb Pain Patients
Brief Title: Novel Non-invasive Brain Stimulation Techniques in Neurological Rehabilitation
Acronym: StimNeuro
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 25C212
Record Dates: First submitted 2023-02-28; First posted 2023-03-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiparesis; Phantom Limb Pain
Keywords: Transcranial Magnetic Stimulation; Paired Associative Stimulation; Stroke; Motor cortex; Phantom limb pain
MeSH Terms: conditions — Stroke; Paresis; Phantom Limb | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: In a first phase [Phase 1], the study aims to assess the motor and neurophysiological effects of a cross-modal 'mirror-PAS' protocol in stroke patients with upper-limb hemiparesis, compared to the standard excitatory M1-PAS.
  In a second phase of the study [Phase 2], we will test the efficacy of the aforementioned cross-modal PAS in a population of amputated patients affected by phantom limb pain (PLP).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [Phase 1] Stroke patients with upper-limb hemiparesis (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation
- [Phase 2] Patients with phantom limb pain (PLP) (Experimental)
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — The standard PAS protocol will be compared with the mirrorPAS protocol.
  Other Names: TMS; Paired associative stimulation

SUMMARY:
Paired associative stimulation (PAS) is a non-invasive brain stimulation protocol, where two stimuli (a peripheral and a cortical one, the latter delivered with transcranial magnetic stimulation - TMS) are repeatedly associated to enhance plasticity in the brain. In the present study, a new cross-modal, visuo-motor PAS protocol - called "mirror-PAS"- will be tested as a possible non-invasive brain stimulation treatment in neurological rehabilitation to promote motor recovery and pain reduction.

Participants will perform the standard PAS targeting the motor system and the recently developed mirror-PAS in two separate sessions. The investigators will compare the possible effect of the protocols in terms of neurophysiological and behavioral outcomes to identify the optimal PAS method to enhance plasticity and promote sensory-motor function.

DETAILED DESCRIPTION:
The motor recovery of the upper limb function, particularly of the hand, is challenging in neurological rehabilitation. Transcranial magnetic stimulation (TMS) is a form of non-invasive brain stimulation that can enhance motor recovery, though promoting brain plasticity of the brain.

In this study, researchers will use a TMS protocol called Paired Associative Stimulation (PAS), in which two stimuli (e.g., a cortical stimulus - delivered with TMS - and a peripheral stimulus) are repeatedly associated to promote associative plasticity in the primary motor cortex (M1).

The objective is to explore the clinical efficacy of a newly developed cross-modal PAS protocol -the so-called "mirror-PAS"- as a possible motor rehabilitation treatment in patients with upper limb motor disorders, investigating its neurophysiological and behavioural effects. The innovative aspect of mirror-PAS is to act on a more extended visuomotor network, featured by the functional properties of the mirror neuron system (MNS). Indeed, in the mirror-PAS, a visual stimulus depicting a hand movement is repeatedly paired with a TMS pulse over M1. In the healthy, this protocol was found effective in modulating neurophysiological responses of the motor cortex (i..e, MEPs), hence inducing these effects bypassing the afferent somatosensory pathway exploited by the standard PAS protocols. This may represent a clinical advantage allowing the promotion of motor recovery through the induction of a plastic reorganization in the damaged motor system by gaining access through a potentially spared MNS.

The project's first phase aims to assess the motor and neurophysiological effects of mirror-PAS in stroke patients with upper-limb hemiparesis, compared to the standard excitatory M1-PAS (whose effects are well known in the literature, even if still debated).

In the second phase, we will test the efficacy of the mirror-PAS in a population of amputated patients affected by phantom limb pain (PLP).

ELIGIBILITY:
Inclusion criteria for stroke patients:

* age from 18 to 85 years
* single, unilateral, hemispheric stroke (cortical or sub-cortical areas)
* stroke confirmed by neuroimaging (CT or MRI)
* stroke at least 4 months before enrollment
* hemiparesis of the upper limb resulting from stroke or hemianesthesia clinically documented

Exclusion criteria for stroke patients:

* contraindications to TMS (Rossi et all, 2021)
* other neurological conditions (e.g., Parkinson's Disease, Multiple Sclerosis, ALS)
* other orthopedic condition that affected the hand (e.g., carpal tunnel syndrome)

Inclusion criteria for PLP patients:

* age from 18 to 90 years
* amputation of one part of the upper limb at least 2 months before enrollment
* presence of stable phantom limb pain at least 2 months prior to enrollment

Exclusion criteria for PLP patients:

* contraindications to TMS (Rossi et all, 2021)
* other neurological, orthopedical or psychiatric conditions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in motor-evoked potentials (MEP) | At baseline and after the administration of the PAS protocols
  [Phase 1, only in stroke patients] peak-to-peak MEP amplitude
Change in functional mapping of phantom limb cortical areas | At baseline and after the administration of the PAS protocols
  [Phase 2, only in PLP patients]

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Bolognini, PhD, Principal Investigator — Laboratorio di Neuropsicologia, IRCCS Istituto Auxologico Italiano
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Lombardy, Italy

REFERENCES:
- [Background] Guidali G, Roncoroni C, Bolognini N. Paired associative stimulations: Novel tools for interacting with sensory and motor cortical plasticity. Behav Brain Res. 2021 Sep 24;414:113484. doi: 10.1016/j.bbr.2021.113484. Epub 2021 Jul 21. PMID 34302877
- [Background] Guidali G, Carneiro MIS, Bolognini N. Paired Associative Stimulation drives the emergence of motor resonance. Brain Stimul. 2020 May-Jun;13(3):627-636. doi: 10.1016/j.brs.2020.01.017. Epub 2020 Feb 5. PMID 32289688
- [Background] Kaur A, Guan Y. Phantom limb pain: A literature review. Chin J Traumatol. 2018 Dec;21(6):366-368. doi: 10.1016/j.cjtee.2018.04.006. Epub 2018 Dec 4. PMID 30583983
- [Background] Castel-Lacanal E, Marque P, Tardy J, de Boissezon X, Guiraud V, Chollet F, Loubinoux I, Moreau MS. Induction of cortical plastic changes in wrist muscles by paired associative stimulation in the recovery phase of stroke patients. Neurorehabil Neural Repair. 2009 May;23(4):366-72. doi: 10.1177/1545968308322841. Epub 2008 Dec 5. PMID 19060132
- [Background] Stefan K, Kunesch E, Cohen LG, Benecke R, Classen J. Induction of plasticity in the human motor cortex by paired associative stimulation. Brain. 2000 Mar;123 Pt 3:572-84. doi: 10.1093/brain/123.3.572. PMID 10686179
- [Background] Hummel FC, Cohen LG. Non-invasive brain stimulation: a new strategy to improve neurorehabilitation after stroke? Lancet Neurol. 2006 Aug;5(8):708-12. doi: 10.1016/S1474-4422(06)70525-7. PMID 16857577
- [Background] Bolognini N, Russo C, Edwards DJ. The sensory side of post-stroke motor rehabilitation. Restor Neurol Neurosci. 2016 Apr 11;34(4):571-86. doi: 10.3233/RNN-150606. PMID 27080070
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615